CLINICAL TRIAL: NCT06943547
Title: The Effectiveness, Cost-effectiveness, and Budget Impact of Interventions to Improve the Delivery of Cervical Cancer Screening in Puerto Rico
Acronym: IMPROVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ana P. Ortiz Martinez, Principal Investigator, University of Puerto Rico Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA282424 (NIH); Protocol #: 2411003902 (Other: IRB - University of Puerto Rico Comprehensive Cancer Center)
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer Screening
Keywords: HPV related cancers; Cervical cancer; Puerto Rico; Patient Navigator; Patient Reminder; HPV self-collection; Cervical cancer prevention; cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A hybrid type 1 effectiveness-implementation study using a four-arm multi-site randomized controlled trial (RCT) conducted within government OBGYN clinics in Puerto Rico. We will assess the effectiveness of patient reminders plus patient navigation and HPV self-collection (individually and in combination) compared to patient reminders alone in increasing cervical cancer screening, timely colposcopy, and cervical precancer treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Patient reminder (Control Arm) (No Intervention): Participants who are due or past recommended cervical cancer screening will be contacted through a scripted telephone call by trained research staff to remind them to schedule an appointment for screening and to provide them with the contact information of the clinic.
- Arm 2: Patient reminder and patient navigator (Experimental): A patient navigator will call the participants to remind them of their cervical cancer screening, assess any screening barriers that they may have, explain the importance of cervical cancer screening, and help them schedule their appointment at the study sites. The patient navigator will also coordinate follow-up colposcopy and treatments as needed.
  Interventions: Behavioral: Arm 2: Patient Navigator
- Arm 3: Patient Reminder and Mailed HPV Test for Self-collection (Experimental): Research staff will contact the participants and remind them to schedule an appointment for cervical cancer screening and will provide them with the contact information of the clinic. She/he will also explain to the participant the role of HPV infection in the development of cervical cancer, provide the participant with information about HPV self-collection, and send them the HPV-self-collection through the mail. The kit will include written instructions on how to collect the cervical sample and mail it back to the study site.
  Interventions: Behavioral: HPV self-collection kit
- Arm 4: Patient reminder, patient navigator, and mailed HPV test for self-collection (Experimental): A patient navigator will remind the participant that it is time for their cervical cancer screening, assess any screening barriers that they may have, explain the importance of cervical cancer screening, and help them schedule their appointment at study sites. She/he will also explain to the participant the role of HPV infection in the development of cervical cancer, provide the participant with information about HPV self-collection, and send them the HPV-self-collection through the mail. The patient navigator will coordinate cytology visits if it is the preference of the participant and any follow-up appointment for cytology and other triage tests, colposcopy and treatments as needed.
  Interventions: Behavioral: Arm 2: Patient Navigator; Behavioral: HPV self-collection kit

INTERVENTIONS:
Behavioral: Arm 2: Patient Navigator — The patient navigation model used in the study is aligned with the conceptual model for cervical cancer screening proposed by the Population-based Research Optimizing Screening Through Personalized Regimens (PROSPR) consortium. The initial contact, as well as most navigation activities, will occur mostly over the phone. In our study, the roles of the patient navigator (Arms 2 and 4) will include: exploring individual barriers to screening, use of motivational interviewing to educate and encourage patients to perform screening, performing reminder calls, and coordinating of referral and clinical services if needed. Also, providing other services to identify and overcome access barriers encountered during the cancer care process, including linkage to community resources. In arm 4, the patient navigator will also facilitate the explanation of the use of the self-collection kits by study participants.
  Arms: Arm 2: Patient reminder and patient navigator; Arm 4: Patient reminder, patient navigator, and mailed HPV test for self-collection
Behavioral: HPV self-collection kit — Each HPV testing kit will include an invitation letter, information sheet, one FLOQSwabs552C® and one sealable plastic bag to put the swab. Because home high risk (HR) HPV self-screening is not standard of care in the US, the kit will also include a letter advising women to receive routine Pap tests, regardless of their HR-HPV self-sampling results. Detailed instructions on how to collect the cervical sample and how to mail the kit back to the study site or bring it to the clinical visit (depending on their preference) will be included.
  Arms: Arm 3: Patient Reminder and Mailed HPV Test for Self-collection; Arm 4: Patient reminder, patient navigator, and mailed HPV test for self-collection

SUMMARY:
Cervical cancer incidence is increasing dramatically (2.5% per year) in Puerto Rico (PR), with increased occurrence of regional (1.7% per year) and distant (4.7% per year) stage cancer, which reflects a real increase and indicates missed screening opportunities. Unfortunately, 80% of cervical cancer cases diagnosed in PR occur among low-income women covered by Medicaid or Medicare, who also have a 70% greater likelihood of being diagnosed with cervical cancer. Cervical cancer screening uptake continues to decline in PR, particularly among low-income Medicaid enrollees, mainly seen by government clinics. Barriers to cervical cancer screening in PR are mainly due to personal (lack of transportation, obesity-related embarrassment) and environmental (repeated disaster events that hampered screening uptake and made recovery slow) factors. The absence of evidence on the effectiveness, cost-effectiveness, and budget impact of patient navigators has limited its adoption among government clinics in this US territory. Multicomponent interventions that can address common screening barriers and improve screening participation in clinic-based settings or avert the need for a clinical-based visit could help improve screening uptake and follow-up care. Our preliminary work suggests the feasibility and acceptability of Human Papillomavirus (HPV) self-sampling in PR. We now propose a hybrid type 1 effectiveness-implementation study using a four-arm multi-site randomized controlled trial (RCT) conducted within government OBGYN clinics in PR. We will assess the effectiveness of patient reminders plus patient navigation and HPV self-collection (individually and in combination) compared to patient reminders alone in increasing cervical cancer screening, timely colposcopy, and cervical precancer treatment (Aim 1). The secondary aim will evaluate key implementation outcomes, including patient and provider receptivity, reach, level of implementation and fidelity, and sustainment intentions. We will then develop an open-cohort micro-simulation model to evaluate the population impact, cost-effectiveness, and budget impact of alternative strategies (Aim 2) to inform their potential applicability at delivery organization, community, and territory levels. This study will provide much-needed knowledge that is necessary to successfully facilitate the adoption and sustained integration of optimal strategies that will improve cervical cancer screening participation and reduce magnifying disparities in Puerto Rico.

DETAILED DESCRIPTION:
Aim 1. Conduct a four-arm multi-site randomized controlled trial to evaluate the effectiveness of three interventions, including patient reminders plus patient navigation and self-collection of HPV test (individually and in combination), compared to patient reminders alone on:

1a. Cervical cancer screening (clinic-based pap test/HPV co-testing) uptake among women and completion of HPV self-collection kit.

1. b. Timely colposcopy and high-grade squamous intraepithelial lesion (HSIL) treatment among women with abnormal screening results. Secondary analyses will examine implementation outcomes, including patient and provider receptivity, reach, level of implementation and fidelity, and sustainment intentions.

   Aim 2. Evaluate the population impact, cost-effectiveness, and budget impact of each intervention strategy compared to patient reminders.
2. a. Develop an open-cohort micro-simulation model of cervical cancer natural history, screening, and treatment outcomes among women in PR and evaluate population impact (incidence and mortality trends) and the cost-effectiveness of alternative strategies.

2b. Evaluate the budget impact of implementing an optimal screening strategy compared to the current intervention mix (at a delivery organization, community, and territory levels).

ELIGIBILITY:
Inclusion Criteria:

* 25-65 years old
* No history of cervical cancer or hysterectomy
* Have not had a Pap test in the past 3 years or more, an HPV test in the past 5 years or more, or a combination of a Pap test and an HPV test in the past 5 or more years (co-testing).
* Must have a record at the study clinics (at least 2 previous visits).

Exclusion Criteria:

* Women with no telephone contact information
* Being pregnant*
* Living with HIV, Lupus, or Crohn's*
* Active on immunotherapy treatment*
* History of organ transplants*

  * Will be excluded as cervical cancer screening guidelines differ for them.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Effectiveness | Within 6 months after a patient is recruited
  Proportion of women who complete cervical cancer screening (attending in-clinic cervical cancer screening) and the proportion of women who completed/returned HPV self-collection kit (Arms 3 and 4).

SECONDARY OUTCOMES:
Screening Adherence after abnormal results | Within 18 months after a patient is recruited.
  Proportion of women who receive a colposcopy after an abnormal Pap Test or positive clinic-based HPV result and the proportion of women who receive treatment after histologically diagnosed HSIL.

OTHER OUTCOMES:
Other tertiary outcomes | Within 18 months after a patient is recruited.
  Revision of the medical record of the participant will permit the evaluation of the following clinical outcomes: Proportion of women with a) abnormal Pap test results, b) cervical high risk HPV infection and c) whose colposcopy results are HSIL/Cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Puerto Rico, San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with research collaborators.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Ortiz AP, Torres-Cintron CR, Santiago-Rodriguez EJ, Ramos-Cartagena JM, Suarez-Ramos T, Damgacioglu H, Colon-Lopez V, Ortiz-Ortiz KJ, Deshmukh AA. Recent cervical cancer incidence, stage at diagnosis, and mortality trends in Puerto Rico, 2001-2019. BMC Med. 2024 Aug 13;22(1):327. doi: 10.1186/s12916-024-03535-4. PMID 39135060